CLINICAL TRIAL: NCT00202410
Title: Phase 2-3 Use of Bacille Calmette-Guèrin (BCG) Vaccine in Patients With a First Clinical Demyelinating Episode: a Multicenter, Randomized, Single Blind Study.
Brief Title: Efficacy of Anti-Tubercular Vaccination in Multiple Sclerosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: S. Andrea Hospital (Other)
Collaborators: Italian Multiple Sclerosis Foundation (Other); Istituto Superiore di Sanità (Other)
Responsible Party: Marco Salvetti, University of Rome "Sapienza"
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEU - BCG - 01
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Tuberculosis vaccine; Therapy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- physiologic solution (Placebo Comparator): subcutaneous administration of physiologic solution
  Interventions: Other: placebo
- Bacille Calmette-Guèrin (BCG) Vaccine (Experimental): Anti-Tubercular Vaccination
  Interventions: Biological: Bacille of Calmette-Guerin

INTERVENTIONS:
Biological: Bacille of Calmette-Guerin — A single intracutaneous dose of 0.1 mL freeze-dried BCG (1 mg/mL; Berna Institute, Basel).
  Arms: Bacille Calmette-Guèrin (BCG) Vaccine
Other: placebo — subcutaneous administration of physiologic solution
  Arms: physiologic solution

SUMMARY:
The frequency of auto-immune diseases (including multiple sclerosis) is increasing in industrialised countries.

According to an hypothesis which is receiving a wide international credit, this may be due to the fact that the populations of these countries are increasingly less exposed to microbes further to the improvement of hygienic conditions and to the use of antibiotics.

If exposure to microbes is lacking, also their regulatory function is missed with a consequent possible onset of auto-immune symptoms.

For this reason, it is deemed that by exposing the immune system of a patient to an ancient microbe, being complex and important in man evolution, like the Tuberculosis Mycobacterium, it is possible to rebalance the immune system.

DETAILED DESCRIPTION:
Vaccination with the Tuberculosis Mycobacterium has proved to be effective in the animal model of multiple sclerosis, experimental allergic encephalitis.

In a study of phase I-II our group has demonstrated the safety of this therapy together with preliminary evidence.

The study includes patients with an initial disease (diagnosis supported by paraclinical criteria): single clinical poly or mono-symptomatic attack in the 6 months preceding the study, MR picture compatible with MS.

Study design 100 randomized patients (i.e. randomly assigned) to be included either in a group of 50 patients undergoing therapy or to a group of 50 patients receiving placebo.

Patients are followed up with monthly contrast MRI for 6 months. At the end of the six months the disease activity in the group of treated patients is benchmarked with the disease activity of the group of patients receiving placebo.

Safety is granted by the extremely wide diffusion of this kind of vaccination worldwide and by the previous study in patients affected by multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an initial disease (diagnosis supported by paraclinical criteria): single clinical poly or mono-symptomatic attack in the 6 months preceding the study, MR picture compatible with MS

Exclusion Criteria:

* Therapy with corticosteroids in the last month
* Plasmapheresis, administration of gamma globulins in the last three months
* Serious heart, renal, hepatic or haematological dysfunction defined by laboratory exams
* Evidence of infections
* Evidence of tubercular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2001-11; Primary Completion 2007-09 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
number of gad-enhancing lesions in T1 | baseline and 6 months
number of lesions in T1 and new lesions in T2 | baseline and 6 months

SECONDARY OUTCOMES:
volume of T2 lesions | 0 and 6 months
volume of T1 lesions (black holes) | 0 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marco Salvetti, Professor, Study Director — S.Andrea Hospital, University of Rome "La Sapienza"; Giovanni Ristori, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Department of Neurology - University of Rome La Sapienza, Rome, Roma, Italy

REFERENCES:
- [Background] Ristori G, Buzzi MG, Sabatini U, Giugni E, Bastianello S, Viselli F, Buttinelli C, Ruggieri S, Colonnese C, Pozzilli C, Salvetti M. Use of Bacille Calmette-Guerin (BCG) in multiple sclerosis. Neurology. 1999 Oct 22;53(7):1588-9. doi: 10.1212/wnl.53.7.1588. PMID 10534275
- [Background] Salvetti M, Pisani A, Bastianello S, Millefiorini E, Buttinelli C, Pozzilli C. Clinical and MRI assessment of disease activity in patients with multiple sclerosis after influenza vaccination. J Neurol. 1995 Feb;242(3):143-6. doi: 10.1007/BF00936886. PMID 7751856
- [Background] Confavreux C, Suissa S, Saddier P, Bourdes V, Vukusic S; Vaccines in Multiple Sclerosis Study Group. Vaccinations and the risk of relapse in multiple sclerosis. Vaccines in Multiple Sclerosis Study Group. N Engl J Med. 2001 Feb 1;344(5):319-26. doi: 10.1056/NEJM200102013440501. PMID 11172162
- [Background] Rook GA, Ristori G, Salvetti M, Giovannoni G, Thompson EJ, Stanford JL. Bacterial vaccines for the treatment of multiple sclerosis and other autoimmune disorders. Immunol Today. 2000 Oct;21(10):503-8. doi: 10.1016/s0167-5699(00)01700-x. No abstract available. PMID 11071529
- [Background] Buttinelli C, Salvetti M, Ristori G. Vaccinations and multiple sclerosis. N Engl J Med. 2001 Jun 7;344(23):1794; author reply 1795-6. No abstract available. PMID 11396455
- [Background] O'Riordan JI, Thompson AJ, Kingsley DP, MacManus DG, Kendall BE, Rudge P, McDonald WI, Miller DH. The prognostic value of brain MRI in clinically isolated syndromes of the CNS. A 10-year follow-up. Brain. 1998 Mar;121 ( Pt 3):495-503. doi: 10.1093/brain/121.3.495. PMID 9549525
- [Background] Brex PA, O'Riordan JI, Miszkiel KA, Moseley IF, Thompson AJ, Plant GT, Miller DH. Multisequence MRI in clinically isolated syndromes and the early development of MS. Neurology. 1999 Oct 12;53(6):1184-90. doi: 10.1212/wnl.53.6.1184. PMID 10522870